CLINICAL TRIAL: NCT01914081
Title: Resveratrol: A Potential Anti- Remodeling Agent in Heart Failure, From Bench to Bedside (RES-HF)
Brief Title: Resveratrol: A Potential Anti- Remodeling Agent in Heart Failure, From Bench to Bedside
Acronym: RES-HF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: Canadian Centre for Agri-Food Research in Health and Medicine (Other); Agriculture and Agri-Food Canada (Other Government); Manitoba Medical Service Foundation (Other)
Responsible Party: Principal Investigator, Dr. Amrit Malik, Cardiologist, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTA/2012/0002; RRC/2011/1169 (Other: St. Boniface Hospital)
Record Dates: First submitted 2013-07-03; First posted 2013-08-01 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; Resveratrol
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resveratrol (Active Comparator): 500 mg (1 capsule BID) of resveratrol for 12 months
  Interventions: Other: Resveratrol
- Placebo (Placebo Comparator): 500 mg (1 capsule BID) of placebo for 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Resveratrol — Patients will receive one uncoated immediate-release caplets containing 500 mg resveratrol, twice daily for the 12 month intervention period
  Other Names: Transmax
  Arms: Resveratrol
Other: Placebo — Patients will receive one uncoated caplet containing placebo, twice daily for the 12 month intervention period
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if resveratrol can improve heart function and quality of life. Although, population studies have revealed that a mild to moderate intake of red wine reduces cardiovascular disease risk in humans, clinical studies that evaluate the potential heart benefits of resveratrol in patients with non-ischemic cardiomyopathy have not been previously reported. Accordingly, this research is being done because it will fill this deficiency in the information available in the literature and establish the clinical benefits of resveratrol in patients with this type of heart disease.

DETAILED DESCRIPTION:
The investigators will conduct a randomized double blinded placebo controlled study of 40 adults (≥18 to 90 years old). Twenty (20) subjects will be included in the placebo arm, and 20 in the treatment arm. Patients will be randomly allocated to receive placebo or resveratrol. After randomization, the two groups of subjects will be followed up in exactly the same way, and the only differences between the care they receive will be those intrinsic to the treatment being compared. The randomization will minimize allocation bias, balancing both known and unknown prognostic factors, in the assignment of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (between 18-90 years of age) with cardiomyopathy, Heart Failure with reduced ejection fraction (HFrEF defined as Left Ventricular Ejection Fraction (LVEF) ≤40%, based on most recent assessment)
* New York Heart Association (NYHA) Functional class II-III (mild-moderate heart failure symptoms)
* On optimal medical management for 6 months as per standard care

Exclusion Criteria:

* Severe valvular cardiomyopathy
* No surgical intervention planned or in past 6 months
* Subjects on \diltiazem (or any other calcium channel blocker)
* Patients with a history of serious hypoglycemia requiring hospitalization or hyperglycemic emergencies requiring hospitalization in the past 6 months
* Subjects on anticoagulants, Coumadin, dabigatran
* Subjects on HIV protease inhibitor (saquinivir), immunosupressants (cyclosporine, tacrolimus)
* Subjects on terfenadine, midazolam, and triazolam
* Subjects on sildenafil or any other drugs used to treat erectile dysfunction
* • Chronic renal failure (defined as estimated glomerular filtration rate (eGFR) ≤30 mL/min per 1.73m2)
* Known liver cirrhosis
* • Other significant comorbidity e.g. cancer affecting ability to complete study
* Pregnant or lactating women
* Subjects on hormone replacement therapy
* Subjects on estrogen containing birth control

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 12 months
  Measured by Minnesota living with heart failure score
Cardiac Function | 12 months
  Echocardiography

SECONDARY OUTCOMES:
Oxidative Stress | 12 Months
  Measurement of oxidative stress using the Oxiselect TBARS Assay.
Total Antioxidant Status | 12 Months
  Measurement of total antioxidant status (TAS) level.
Inflammatory Marker Measurements | 12 Months
  Inflammatory markers will be measured by plasma levels of interleukin 6 (IL6) and tumor necrosis factor (TNF).
Nitric Oxide Determination | 12 Months
  Total nitric oxide levels will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Zieroth, MD, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No